CLINICAL TRIAL: NCT02537444
Title: A Phase 2 Proof-of-Concept Study of ACP-196 Alone and in Combination With Pembrolizumab in Subjects With Recurrent Ovarian Cancer
Brief Title: Acalabrutinib (ACP-196) Alone and in Combination With Pembrolizumab in Ovarian Cancer (KEYNOTE191)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-208
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — acalabrutinib

ARMS (2):
- Regimen 1 (Experimental): Drug: acalabrutinib monotherapy
  Interventions: Drug: Acalabrutinib
- Regimen 2 (Experimental): Drug: Combination of acalabrutinib and pembrolizumab
  Interventions: Drug: acalabrutinib and pembrolizumab combination

INTERVENTIONS:
Drug: Acalabrutinib
  Other Names: ACP-196
  Arms: Regimen 1
Drug: acalabrutinib and pembrolizumab combination
  Arms: Regimen 2

SUMMARY:
To characterize the safety and efficacy of acalabrutinib (ACP-196) monotherapy and acalabrutinib plus pembrolizumab combination therapy in subjects with recurrent ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age.
* Histologically confirmed ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma.
* Progression of disease after the most recent anticancer treatment. At least 1 prior chemotherapy regimen must have included a taxane.
* Platinum-sensitive ovarian cancer defined by recurrence or progression of disease > 6 AND < 24 months after completion of the most recent platinum-based therapy.
* Measurable disease as defined by RECIST 1.1.
* ECOG performance status of 0 or 1.
* Completion of all therapy for the treatment of cancer 2 weeks before the start of study therapy and recovered.

Exclusion Criteria:

* Evidence of platinum-refractory ovarian cancer defined as recurrence or progression during the first 6 cycles of or < 6 months after the beginning of first-line platinum based chemotherapy.
* Evidence of platinum-resistant ovarian cancer defined as recurrence or progression within 6 months after completing the most recent platinum-based therapy.
* More than 3 prior lines of cytotoxic chemotherapy for ovarian cancer.
* Prior malignancy (other than ovarian cancer), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years.
* Breastfeeding and pregnant.
* Known central nervous system metastases and/or carcinomatous meningitis.
* Subjects with active cardiovascular disease not medically controlled or those who have had myocardial infarction in the past 6 months..
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (2):
- United States (2):
  - Arizona Gynecology Oncology, Tucson, Arizona
  - Jordan Center For Gynecologic Cancer At Penn, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Acalabrutinib Monotherapy: Acalabrutinib 100mg administered orally (PO) twice daily BID.
- Arm 2 - Acalabrutinib + Pembrolizumab: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
Started | 39 | 39
Enrolled | 39 | 39
Received Study Medication | 38 | 39
Discontinued Study | 39 | 39
Completed | 0 | 0
Not Completed | 39 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (11.52) | 64.2 (12.75) | 64.4 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 12 weeks for up to 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 - Acalabrutinib Monotherapy: Acalabrutinib 100mg administered orally (PO) twice daily.
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 35 | 33
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Safety Analysis tracked from 0 day to 2 years.
Groups:
- Arm 1 - Acalabrutinib Monotherapy: Acalabrutinib 100mg administered orally (PO) twice daily (BID).
- Arm 2 - Acalabrutinib + Pembrolizumab: Acalabrutinib 100mg plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 16/38 | 22/39
Serious Adverse Events (participants affected / at risk) | 8/38 | 16/39
Other Adverse Events (participants affected / at risk) | 34/38 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Acalabrutinib Monotherapy (N=38) | Arm 2 - Acalabrutinib + Pembrolizumab (N=39)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 5
Ascites (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1 — General Disorders and Administration Site Conditions
Non-Cardiac Chest Pain (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 1 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Acalabrutinib Monotherapy (N=38) | Arm 2 - Acalabrutinib + Pembrolizumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Sinus Tachycardia (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Vision Blurred (Eye disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 16 | 29
Diarrhea (Gastrointestinal disorders) | 17 | 11
Vomiting (Gastrointestinal disorders) | 7 | 21
Abdominal Pain (Gastrointestinal disorders) | 9 | 14
Abdominal Distension (Gastrointestinal disorders) | 7 | 6
Constipation (Gastrointestinal disorders) | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 2 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 16 | 20 — General Disorders and Administration Site Conditions
Oedema Peripheral (General disorders) | 3 | 4 — General Disorders and Administration Site Conditions
Chills (General disorders) | 4 | 5 — General Disorders and Administration Site Conditions
Pyrexia (General disorders) | 2 | 5 — General Disorders and Administration Site Conditions
Pain (General disorders) | 1 | 2 — General Disorders and Administration Site Conditions
Non-Cardiac Chest Pain (General disorders) | 2 | 1 — General Disorders and Administration Site Conditions
Urinary Tract Infection (Infections and infestations) | 5 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 8 | 6
Alanine Aminotransferase Increased (Investigations) | 4 | 10
Aspartate Aminotransferase Increased (Investigations) | 4 | 9
Blood Creatinine Increased (Investigations) | 2 | 3
Weight Decreased (Investigations) | 1 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 3
Lymphocyte Count Decreased (Investigations) | 1 | 3
Platelet Count Decreased (Investigations) | 0 | 3
White Blood Cell Count Decreased (Investigations) | 0 | 4
Breath Sounds Abnormal (Investigations) | 0 | 3
Protein Total Decreased (Investigations) | 0 | 3
Carbohydrate Antigen 125 Increased (Investigations) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 10
Dehydration (Metabolism and nutrition disorders) | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Musculoskeletel Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 17 | 21
Neuropathy Peripheral (Nervous system disorders) | 2 | 4
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 7
Depression (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Vaginal Haematuria (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 7
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hot Flush (Vascular disorders) | 2 | 3
Dizziness (Nervous system disorders) | 9 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02537444/SAP_000.pdf
  • Study Protocol (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT02537444/Prot_001.pdf